CLINICAL TRIAL: NCT03620799
Title: Effectiveness of a Roller Intervention in Patients With Anterior Knee Pain: a Randomized Controlled Trial
Brief Title: Efffectiveness of a Roller Intervention in Anterior Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DF0076UG
Record Dates: First submitted 2018-07-24; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Roller intervention; Knee pain; Algometry
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 10 participants will be assigned to the intervention group in order to the inclusion criteria for the study. Experimental group. Manual therapy intervention
  Interventions: Procedure: Manual therapy
- Control group (No Intervention): 10 participants will be assigned to the control group in order to the inclusion criteria for the study. Control group

INTERVENTIONS:
Procedure: Manual therapy — A manual intervention technique is employed to the intervention group based on a roller treatment.
  Arms: Intervention group

SUMMARY:
Anterior knee pain is one of the most frequent reasons for consultation within knee conditions in adolescents and young adults. However, despite the high prevalence of this disorder, its pathogenesis and therefore its treatment are not clearly understood. Foam rolling has become a common intervention to enhance joint mobility and muscle recovery after exercise. the aim of this study is analyze the effectiveness of a roller intervention in patients with anterior knee pain.

DETAILED DESCRIPTION:
Randomized controlled trial. patients were divided into two groups, intervention and control.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years.
* Knee anterior pain diagnosis

Exclusion Criteria:

* Concomitant somatic or psychiatric disorder
* Previous knee surgery
* Other lower limb traumatological pathologies

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2018-09-10 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in mechanosensitivity | Changes from baseline mechanosensitivity at 4 weeks
  Mechanosensitivity is going to be assessed by a hand-held pressure algometer. The pressure will be applied perpendicular to the skin at a constant rate of 30 kPa/s until the patient felt the pressure change to pain and pressed a button defining the PPT.

SECONDARY OUTCOMES:
Vertical jump assessment with a mat | Baseline, 4 weeks
  The subject started with the foot of the designated testing leg on the contact mat and their hands on their hips, they were then instructed to sink and hold a knee position (approximately 1208 knee angle), and the experimenter then counted out 4 s. On the count of four the subject was instructed to then jump as high as possible.
Isokinetic strength | Baseline, 4 weeks
  Isokinetic strength of the knee flexors and extensors of each leg will be measured using an isokinetic Biodex dynamometer (Biodex Corporation, Shirley, NY), which recorded instantaneous muscular torques.
Pain intensity assessed by the Brief Pain Inventory | Baseline, 4 weeks
  Pain will be assessed using the Brief Pain Inventory. The Brief Pain Inventory is a pain assessment tool used to measure pain intensity and pain interference. Patients rate the severity of their pain at its worst and least during the previous week, on average, and "right now". Patients rate their level of pain interference in different contexts.
Functional knee limitation assessed by the Kujala Knee Score | Baseline, 4 weeks
  The Kujala Knee Score questionnaire will be selected for self-reported functional activity level of the patients. The composite score ranges from 0 to 100, with 100 indicating no functional limitation.

IPD SHARING:
Plan to Share IPD: Undecided